CLINICAL TRIAL: NCT06326112
Title: Role of Active Deresuscitation After Resuscitation: The RADAR-Canada Pilot Clinical Trial
Brief Title: Role of Active Deresuscitation After Resuscitation:
Acronym: RADAR-Canada
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, John Marshall, Professor of Surgery and Critical Care Medicine, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4588
Record Dates: First submitted 2024-02-26; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Fluid Overload; Critical Illness; Sepsis; ARDS; Trauma
Keywords: sepsis; acute respiratory distress syndrome; multiple trauma; critical illness
MeSH Terms: conditions — Edema; Critical Illness; Sepsis; Wounds and Injuries; Respiratory Distress Syndrome; Multiple Trauma | interventions — Furosemide; Metolazone

STUDY DESIGN:
Intervention Model Description: RADAR-Canada is a parallel group CT in which study participants are randomized in a 1:1 ratio to protocolized deresuscitation or usual care
Who Masked: Outcomes Assessor
Masking Description: Masking of the health care team will not be feasible as they must administer the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active deresuscitation (Experimental): * Fluid minimization: clinical and research teams will review all intravenous orders and attempt to reduce fluids to 10-15 ml/hr.
  * Active deresuscitation:
  * Administer bolus furosemide 0.5 mg/kg bid or tid
  * Target daily negative fluid balance as follows:
  Calculated positive balance:
  < 3 liters -600 - -800 ml/24 hours 3-6 liters 0.8 - 1.2 liters/24 hours 6- 10 liters 1.2 - 2.0 liters/24 hours >10 liters >2.0 liters/24 hours
  * If bolus furosemide fails to achieve these goals, results in hypotension or tachycardia, or at the discretion of the attending intensivist, start furosemide infusion titrated on an hourly basis to achieve above goals
  * If single agent ineffective, consider addition of metolazone
  Interventions: Drug: Furosemide Injection; Drug: Metolazone Tablets
- Usual care (No Intervention): Care at the discretion of the attending team.

INTERVENTIONS:
Drug: Furosemide Injection — o.5 mg/kg bid or tid IV
  Arms: Active deresuscitation
Drug: Metolazone Tablets — Diuretic as needed
  Arms: Active deresuscitation

SUMMARY:
The RADAR-Canada trial is a pilot RCT undertaken to assess the acceptability of, compliance with, and biologic consequences of a deresuscitation protocol designed to expedite the removal of excess interstitial fluid in patients who remain in a positive fluid balance following admission to an intensive care unit (ICU).

DETAILED DESCRIPTION:
Background: Over the course of an acute illness, critically ill patients typically receive substantial volumes of intravenous fluids, administered for resuscitation, maintenance, and as diluents for medications. A positive fluid balance is associated with adverse clinical outcomes. Whether active reversal of a positive fluid balance through fluid restriction and diuresis will improve outcomes is uncertain.

Methods: The Role of Active Deresuscitation After Resuscitation (RADAR) trial is a pilot study to determine the feasibility of a larger trial powered for clinically important outcomes, the acceptability of a deresuscitation protocol, and the impact of a trial on stability of practice patterns. RADAR is an open label pilot trial that will recruit 120 patients from 10 to 12 active sites in Canada. Eligible patients will be 18 years or older, mechanically ventilated >48 hours but in the ICU for less than five days, and in a calculated positive fluid balance of > three liters. Patients will be randomized to either usual care or a deresuscitation protocol incorporating a fluid minimization strategy and diuresis.

Results and Discussion: Evidence that recruited patients will be managed according to the trial protocol, with a withdrawal rate of less than 5%, a compliance rate of >75% and a crossover rate of <10% will establish the acceptability of the protocol. A mean difference in fluid balance between groups of more than three liters 72 hours after enrolment will establish the feasibility of the protocol. Analyses of clinical effects will be secondary analyses. Survival to day 90 following randomization will be measured, and other clinical measures will provide estimates of rates of key outcomes to inform the design of a definitive, adequately powered trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Mechanically ventilated for > 48 hours
3. Calculated volume accumulation > 3 liters since ICU admission or pitting edema in at least two sites (arms, legs, or trunk)
4. Admitted to ICU for ≤ five days
5. Informed consent obtained from patient or alternate decision-maker

Exclusion Criteria:

1. Lack of consent from patient or substitute decision maker or from responsible physician 2. Active bleeding (defined as > 2 units transfused RBC in past 24 hours) 3. Hemodynamic instability (defined as use of vasopressors >0.1 µg/kg/minute norepinephrine or equivalent, or increase in vasopressor dose over past 6 hours) 4. Currently receiving dialysis, or plans to initiate dialysis imminently 5. P/F ratio < 75 6. Subarachnoid hemorrhage 7. Severe traumatic brain injury with admission GCS <8 8. Diabetic ketoacidosis or hyperosmolar state 9. Acute cardiac failure or cardiogenic shock 10. Suspected or established diabetes insipidus 11. Allergy to furosemide 12. High probability of death within 24 hours

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Mean cumulative fluid balance | 72 hours following randomization
  Total fluid input (mL) - output (mL) in each group
Compliance with deresuscitation protocol | Each 24 hours over first week
  Daily fluid balance in mL >10 liters, target >2.0 liters/24 hours
Acceptability of protocol | Day 1
  Percentage of eligible patients who consent to randomization

SECONDARY OUTCOMES:
All cause mortality | 90 days following randomization
  Deaths
New onset organ dysfunction | 7 days following randomization
  Change in aggregate Multiple Organ Dysfunction (MOD) score from baseline, where the range is 0 - 25, and higher values indicate more severe organ dysfunction
Organ support-free days | 28 days following randomization
  Days alive and free from respiratory or hemodynamic support

OTHER OUTCOMES:
Inflammatory and renal biomarkers - change from baseline values | 3 days following randomization
  including, but not limited to IL-6, sTNFr1, ICAM, HCO3-, protein C, CRP) or markers of AKI (including, but not limited to N-GAL, KIM-1, TIMP2-IGFBP-7, cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: John C Marshall, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada